CLINICAL TRIAL: NCT06423118
Title: Cross-sectional Investigation of Sleep Apnea and Cognition in Older Adults Using the ANNE Vital Sign System
Brief Title: Sleep Apnea and Cognition in Older Adults
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Alzheimer Society of Canada (Other)
Responsible Party: Principal Investigator, Dr. Jennifer Rabin, Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 5140
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Sleep; Cognition; Aging
Keywords: sleep; cognition; aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Healthy Older Adults: * Age 55-85
  * 8+ years of education
  * No frank cognitive impairment or dementia
  Interventions: Device: ANNE Vital Sign System

INTERVENTIONS:
Device: ANNE Vital Sign System — The ANNE Vital Sign System is a pair of non-invasive, flexible sensors originally designed for vital signs monitoring in the paediatric intensive care unit.
  Other Names: ANNE One

SUMMARY:
The goal of this cross-sectional, observational, medical device trial is to examine the association of several sleep parameters, including specific respiratory events and an apnea-hypopnea index, with cognitive performance in older adults. The main question the study aims to answer is:

Is there an association between sleep parameters with cognitive performance?

Researchers will collect sleep parameters from participants using a device called the ANNE Vital Sign System and will test whether they are associated with performance on different memory and thinking tasks.

Participants will:

Complete a battery of cognitive tests to assess their memory and thinking performance.

Wear the ANNE Vital Sign System continuously for a period of 24 hours.

DETAILED DESCRIPTION:
Nearly a third of older adults experience difficulty initiating or maintaining sleep and nearly half have sleep apnea. However, current reliance on gold-standard in-lab polysomnography has been a barrier to detecting, quantifying, and measuring these sleep problems. Polysomnography is difficult for many older adults to tolerate, requires specialized technologists to obtain and analyze the recordings, is labour intensive and expensive, and not widely available in many jurisdictions, all of which impede use by primary care clinicians or end-users. Recent advances in wearable sensor development have led to a new generation of wearable sensors that have good potential to overcome these barriers.

Accumulating evidence suggests that poor sleep quality increases the risk of cognitive impairment and dementia, however studies in older adults linking objectively measured sleep function with comprehensive cognitive testing are lacking. The primary objective of this cross-sectional study is to examine the association of several objectively measured sleep parameters (e.g., sleep apnea) with cognitive performance.

The Advanced NeoNatal Epidermal (ANNE) Vital Sign System was created for the purposes of providing real-time vital signs monitoring in the paediatric intensive care unit. The ANNE Vital Sign System integrates simultaneous synchronized ambulatory measurement of electrocardiography, photoplethysmography with derived pulse oximetry, pulse arrival time with derived beat-to-beat blood pressure, triaxial accelerometry, respiratory rate, and temperature, to enable accurate measurement of sleep apnea. The characteristics that make the ANNE Vital Sign System ideal for use in children (non-invasive, flexible, ease of use, comfort, skin safety) also make it ideal for use in adults. Compelling in-laboratory preliminary data from our collaborator at Sunnybrook Research Institute (SRI) has demonstrated the capacity for ANNE to detect and characterize sleep apnea in older adults.

After the informed consent process, participants will complete a 1-hour battery of cognitive tests. If participants have completed the same set of cognitive tests in the past year at SRI no cognitive testing will take place.

Following testing, participants will be shown how to affix and remove the sensors to their chest and dominant index finger (or non-dominant if dominant is not available) according to manufacturer recommendations. Participants will be given the device to take home and asked to wear the sensors for a 24-hour period. They will also be provided with ANNE chest adhesive, ANNE limb adhesive, and a clinical waterproof 3M Tegaderm dressing. Participation in the study concludes after the device is worn for the 24-hour period.

Though there are no substantial benefits for participants, this study may lead to a better understanding of the association between sleep apnea and cognition in older adults. Given that poor sleep quality is a risk factor for dementia, there is a need to better characterize the relationship between objective sleep parameters and cognition.

ELIGIBILITY:
Inclusion Criteria:

1. Sufficient knowledge of English to understand and provide informed consent
2. Competent to provide consent
3. Aged 55-85, Male and Female
4. ≥ 8 years of education
5. Capable of cooperating for the duration of the study procedures and assessments
6. No frank cognitive impairment or dementia
7. Sufficient (corrected) vision to participate in cognitive testing
8. Sufficient (corrected) hearing to participate in cognitive testing

Exclusion Criteria:

1. Cannot read and comprehend English language instructions
2. Major cardio- or cerebro-vascular event (heart attack, stroke, significant white matter changes)
3. Unstable diseases (e.g., pulmonary, endocrine disorder)
4. Active malignancy or infectious diseases
5. History of significant learning disability
6. Major psychiatric/neurologic/degenerative disorder, including a diagnosis of mild cognitive impairment or dementia
7. History of significant head trauma or recurrent concussions requiring hospitalization followed by persistent neurologic defaults or known structural brain abnormalities
8. Pain or sleep disorder that could interfere with cognitive testing
9. Major medical concerns that might interfere with cognitive testing
10. Recent history of substance/drug abuse
11. Known nickel allergy
12. Known cardiac implantable device
13. Known arrhythmias
14. Outside the included age range
15. Pregnant or breast feeding
16. Otherwise unable to use the ANNE sensors; for example, finger amputations.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy older adults between the ages of 55-85, with 8+ years of education and no frank cognitive impairment or dementia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2034-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Association between apnea-hypopnea index and cognitive performance | 24 hours
  An apnea-hypopnea index, the combined average number of apneas and hypopneas that occur per hour of sleep, will be calculated from ANNE Vital Sign System data. Study staff will annotate apneas and hypopneas to calculate the index using an EEG annotation tool.
  A linear regression model will be constructed to examine the association between apnea-hypopnea index and performance on a battery of neuropsychological tests, which includes:
  1. Montreal Cognitive Assessment
  2. Free and Cued Selective Reminding Test
  3. Benson Complex Figure Copy
  4. Doors Test, Parts A and B
  5. WAIS-III Symbol Digit Coding
  6. Benson Complex Figure Delay
  7. Benson Complex Figure Recognition
  8. 7-24 Spatial Recall Test
  9. Colour Trails Test, parts 1 and 2
  10. Controlled Oral Word Association Test (FAS)
  11. Semantic Fluency (Animals)
  12. Trail Making Test, parts A and B

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rabin, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foley DJ, Monjan AA, Brown SL, Simonsick EM, Wallace RB, Blazer DG. Sleep complaints among elderly persons: an epidemiologic study of three communities. Sleep. 1995 Jul;18(6):425-32. doi: 10.1093/sleep/18.6.425. PMID 7481413
- [Background] Senaratna CV, Perret JL, Lodge CJ, Lowe AJ, Campbell BE, Matheson MC, Hamilton GS, Dharmage SC. Prevalence of obstructive sleep apnea in the general population: A systematic review. Sleep Med Rev. 2017 Aug;34:70-81. doi: 10.1016/j.smrv.2016.07.002. Epub 2016 Jul 18. PMID 27568340
- [Background] Oosterman JM, van Someren EJ, Vogels RL, Van Harten B, Scherder EJ. Fragmentation of the rest-activity rhythm correlates with age-related cognitive deficits. J Sleep Res. 2009 Mar;18(1):129-35. doi: 10.1111/j.1365-2869.2008.00704.x. PMID 19250179
- [Background] Shi L, Chen SJ, Ma MY, Bao YP, Han Y, Wang YM, Shi J, Vitiello MV, Lu L. Sleep disturbances increase the risk of dementia: A systematic review and meta-analysis. Sleep Med Rev. 2018 Aug;40:4-16. doi: 10.1016/j.smrv.2017.06.010. Epub 2017 Jul 6. PMID 28890168
- [Background] Sindi S, Kareholt I, Johansson L, Skoog J, Sjoberg L, Wang HX, Johansson B, Fratiglioni L, Soininen H, Solomon A, Skoog I, Kivipelto M. Sleep disturbances and dementia risk: A multicenter study. Alzheimers Dement. 2018 Oct;14(10):1235-1242. doi: 10.1016/j.jalz.2018.05.012. Epub 2018 Jul 17. PMID 30030112
- [Background] Zhu X, Zhao Y. Sleep-disordered breathing and the risk of cognitive decline: a meta-analysis of 19,940 participants. Sleep Breath. 2018 Mar;22(1):165-173. doi: 10.1007/s11325-017-1562-x. Epub 2017 Sep 13. PMID 28905231
- [Background] Chung HU, Kim BH, Lee JY, Lee J, Xie Z, Ibler EM, Lee K, Banks A, Jeong JY, Kim J, Ogle C, Grande D, Yu Y, Jang H, Assem P, Ryu D, Kwak JW, Namkoong M, Park JB, Lee Y, Kim DH, Ryu A, Jeong J, You K, Ji B, Liu Z, Huo Q, Feng X, Deng Y, Xu Y, Jang KI, Kim J, Zhang Y, Ghaffari R, Rand CM, Schau M, Hamvas A, Weese-Mayer DE, Huang Y, Lee SM, Lee CH, Shanbhag NR, Paller AS, Xu S, Rogers JA. Binodal, wireless epidermal electronic systems with in-sensor analytics for neonatal intensive care. Science. 2019 Mar 1;363(6430):eaau0780. doi: 10.1126/science.aau0780. PMID 30819934

DOCUMENTS (1):
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT06423118/ICF_000.pdf